CLINICAL TRIAL: NCT01073722
Title: Endobronchial EZ Blocker Compared to Left Sided Double-lumen Tube for One-lung Ventilation
Brief Title: EZ Blocker Versus Left Sided Double-lumen Tube
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Dr. J.M.J. Mourisse, Radboud University Nijmegen Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL30799,091,09
Record Dates: First submitted 2010-02-17; First posted 2010-02-23 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2010-08

CONDITIONS: One-lung Ventilation
Keywords: thoracic surgery; one-lung ventilation; double lumen tube; endobronchial blocker
MeSH Terms: interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Left double lumen tube (Active Comparator): Traditionally, single lung ventilation is obtained with a double lumen tube (DLT). In our institution a polyvinyl DLT (Broncho-cath, Mallinckrodt,) without carinal hook, is used. This type of tube exists of a tube with two lumen with two distal cuffs. One lumen (called the bronchial lumen) extends some distance further, has a slight curvature and has a small blue cuff. The other lumen (called the tracheal lumen) has a larger cuff. A DLT tube exists in four sizes and one can choose in a left or a right configuration. Almost always, we use a left sided DLT. A DLT has a much larger diameter than a standard single lumen endotracheal tube
  Interventions: Device: Placement of double lumen tube for one-lung ventilation
- EZ-blocker (Active Comparator): The EZ-blocker (EZB) is a semi-rigid catheter but it has two distal extensions, both with an inflatable cuff and a central lumen. It is intended for use in combination with a standard single lumen tube. After the EZB is advanced trough the distal end of the single lumen tube, both extensions spread out and find their way in the left and right main stem bronchi. The place where the two extensions are attached to the shaft now rests on the carina. Fiber optic bronchoscopy should be used for proper positioning. After placement of the EZB, one of the cuffs can be inflated to obtain lung separation under direct visual inspection with fiber optic bronchoscopy.
  Interventions: Device: Placement of EZ- Blocker for one-lung ventilation

INTERVENTIONS:
Device: Placement of double lumen tube for one-lung ventilation — The gold standard for lung isolation is the use of a double lumen tube (DLT). A DLT is a bifurcated tube with a bronchial and a tracheal lumen.
  Other Names: Broncho-cath (Mallinckrodt)
  Arms: Left double lumen tube
Device: Placement of EZ- Blocker for one-lung ventilation — Bronchial blockers are balloon-tipped semi-rigid catheters. Different types are available. They are not easy to put in position and frequently dislocates during repositioning of the patient or during surgical manipulation. To solve these problems, a novel type of bronchus blocker, i.e. the EZ- Blocker® is developed. The EZB is also a semi-rigid catheter but it has two distal extensions, both with an inflatable cuff and a central lumen. These improvements owe to the fact that the blocker anchors itself on the carina with the two extensions.
  Other Names: EZ-blocker (AnaesthetIQ BV, Rotterdam, The Netherlands)
  Arms: EZ-blocker

SUMMARY:
Lung isolation is used to achieve one lung ventilation to facilitate thoracic surgery. Two methods are commonly used, a double lumen tube (DLT) or a bronchial blocker introduced through a single lumen tube. However, both techniques have advantages and disadvantages. Briefly, the DLT can be positioned faster and remains firmly in place, but is sometimes difficult or even impossible to introduce. The DLT is larger than a conventional single lumen tube and the incidence of postoperative hoarseness and airway injuries is higher. Compared to the DLT, bronchial blocking devices are more difficult to position and need more frequent intraoperative repositioning. These disadvantages of the existing devices for lung isolation prompted further development of the bronchial blocker concept. The design of a new Y shaped bronchial blocker, the EZ- Blocker® (AnaesthetIQ BV, Rotterdam, The Netherlands) (EZB), combines the advantages of both lung isolation techniques. The aim of the study is to compare in a randomised, prospective way the ease of placement, the incidence of malpositioning and the quality of lung deflation of a left DLT and a EZB. Secondly, the incidence and severity of damage to laryngeal, tracheal and bronchial structures caused by the use of the DLT or the EZB is a target of the study.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3 patients
* Patients scheduled for surgery requiring a left sided DLT for single lung ventilation

Exclusion Criteria:

* Contraindications are lesions along the path of the left sided double lumen tube or the EZB
* Tracheal or mainstem bronchial stenosis
* Distorted carinal anatomy,
* Anticipated difficult intubation (Mallampatti score ≥ 3)
* History or presence of tracheostoma
* Patients who require absolute lung separation
* Patients who require sleeve resection of mainstem bronchus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
the incidence of malposition of a left sided DLT or the EZB | there are four time points (after insertion of the device, after inflation of cuff or balloon, after repositioning patient, during surgery) were malposition are considered. Total time spend is 3 hours on the day of the operation

SECONDARY OUTCOMES:
description of damage to laryngeal, tracheal and bronchial structures | videobronchoscopy before and after intervention. Time frame 5 min for each video and additional 5 min for assessment afterwards on the day of the operation
the ease of insertion | the ease of insertion of the devices is qualitative variable: 1= excellent, 2= good, 3=average, 4=poor. Time frame is 5 min on the day of the operation.
the incidence of postoperative complains of sore throat and hoarseness | questionnaire (2 questions, time frame is 1 min) after surgery and one day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jo Mourisse, Dr., Principal Investigator — Department of anesthesiology, pain and palliative medicine of the Radboud University Nijmegen Medial Center
Locations (1):
- Department of Anesthesiology, Pain and Palliative Medicine of the Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands